CLINICAL TRIAL: NCT04678674
Title: Autogenous Tooth Roots for Lateral Alveolar Ridge Augmentation and Staged Implant Placement
Brief Title: Tooth Roots for Lateral Alveolar Ridge Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Catherine Specialty Hospital (Other)
Responsible Party: Principal Investigator, Igor Smojver, Principal Investigator, St. Catherine Specialty Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16041985
Record Dates: First submitted 2020-12-08; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Bone Atrophy, Alveolar
Keywords: bone augmentation; autogenous tooth roots; dental implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone defect surgery (Experimental): augmentation on insufficient alveolar ridges with autologous teeth will be performed (wisdom tooth or periodontally compromised tooth)
  Interventions: Procedure: tooth root augmentation

INTERVENTIONS:
Procedure: tooth root augmentation — Autogenous tooth roots for lateral alveolar ridge augmentation and staged implant placement.

SUMMARY:
A deficient alveolar ridge segment in prepara¬tion for implant placement can be regenerated by several techniques. The type of graft material for each patient depends on many factors such as the anatomy, the morphology of the bone defect, type of prosthodontic rehabilitation and patient or clinician preferences. Bone graft material should have three properties that made it ideal: a) osteoconduction, it provides scaffolds for bone regeneration; b) osteoinduction, it promotes the recruitment of bone-forming cells and formation of bone and c) osteogenesis, induction of cells in the graft to promote regeneration of the bone.

Despite of the development of different types of graft material, autogenous bone is still the gold standard for bone augmentation because it exhibits these three mentioned properties. Although it has many advantages, autologous bone has some disadvantages such as high resorption rate up to 50 %, limited source and donor site morbidity. Allografts, xenografts and alloplastic bone graft are materials that are used in everyday practice and over long period, but their disadvantages are numerous in comparison with autologous bone. Allografts can be carrier of some disease and show lack of osteoproliferation, while alloplasts and xenografts show only osteoconduction. According to these facts, it is obvious that there is a need for development an alternative graft material that will surpass these disadvantages.The reconstruction of deficient alveolar ridge defect by the lateral bone augmentation prior to the dental implant placement is predictable and commonly used method. Except animal studies, recent clinical studies showed that there is no difference in the osseointegration of titanium implants in deficient alveolar ridges reconstructed with autogenous cortical bone blocks or autogenous teeth.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 years
* candidate for lateral ridge augmentation
* insufficient bone ridge width at the recipient site for implant placement
* sufficient bone height at the recipient site for implant placement and (e)
* healthy oral mucosa
* at least 2 mm keratinized tissue

Exclusion Criteria:

* general contraindications for dental and/or surgical treatments
* inflammatory and autoimmune disease of the oral cavity,
* uncontrolled diabetes (HbA1c > 7%)
* history of chemotherapy or radiotherapy within the past five years,
* previous immunosuppressant, bisphosphonate or high- dose corticosteroid therapy
* smokers
* pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was defined as the clinical width (CW) of the alveolar ridge | 6 months
  The primary endpoint was defined as the clinical width (CW) of the alveolar ridge being sufficient for the placement of an adequately dimensioned dental implant without the need for a secondary grafting at 6 months after surgery in either group. CW was assessed before (CWa) and after (CWb) augmentation healing period of 6 months in cone-beam computed tomography (CBCT) scans.
  Measurements were performed to the nearest 0.5mm below the crest using a CBCT.

SECONDARY OUTCOMES:
Periimplant tissue stability of augmented sites after prosthetic rehabilitation | 12 months
  Usage of periimplant tissue parameters for assessing the conditions around implants placed in augmented sites using pink esthetic score (PES) that evaluates the esthetic outcome of soft tissue around implant-supported single crowns by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency.
gain in ridge width (CWg) | 6 months
  CWg (mm) = CWb ( ridge after surgery in mm)- CWa ( ridge before surgery in mm)
soft tissue dehiscences | 6 months
  yes/no for secondary wound healing
wound infections | 6 months
  monitoring whether there is an increased incidence of inflammatory conditions after the specified procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Gabrić, PhD, Study Director — School of Dental Medicine Zagreb
Locations (1):
- St. Catherine Specialty Hospital, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
individual participant data will be available all time
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 moths
Access Criteria: only researchers

REFERENCES:
- [Background] Misch CM, Jensen OT, Pikos MA, Malmquist JP. Vertical bone augmentation using recombinant bone morphogenetic protein, mineralized bone allograft, and titanium mesh: a retrospective cone beam computed tomography study. Int J Oral Maxillofac Implants. 2015 Jan-Feb;30(1):202-7. doi: 10.11607/jomi.3977. PMID 25615925
- [Background] Roccuzzo M, Ramieri G, Bunino M, Berrone S. Autogenous bone graft alone or associated with titanium mesh for vertical alveolar ridge augmentation: a controlled clinical trial. Clin Oral Implants Res. 2007 Jun;18(3):286-94. doi: 10.1111/j.1600-0501.2006.01301.x. Epub 2007 Feb 13. PMID 17298495
- [Background] Naenni N, Lim HC, Papageorgiou SN, Hammerle CHF. Efficacy of lateral bone augmentation prior to implant placement: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:287-306. doi: 10.1111/jcpe.13052. PMID 30624791
- [Result] Nampo T, Watahiki J, Enomoto A, Taguchi T, Ono M, Nakano H, Yamamoto G, Irie T, Tachikawa T, Maki K. A new method for alveolar bone repair using extracted teeth for the graft material. J Periodontol. 2010 Sep;81(9):1264-72. doi: 10.1902/jop.2010.100016. PMID 20476887
- [Result] Qin X, Raj RM, Liao XF, Shi W, Ma B, Gong SQ, Chen WM, Zhou B. Using rigidly fixed autogenous tooth graft to repair bone defect: an animal model. Dent Traumatol. 2014 Oct;30(5):380-384. doi: 10.1111/edt.12101. Epub 2014 Mar 5. PMID 24597718
- [Result] Becker K, Drescher D, Honscheid R, Golubovic V, Mihatovic I, Schwarz F. Biomechanical, micro-computed tomographic and immunohistochemical analysis of early osseous integration at titanium implants placed following lateral ridge augmentation using extracted tooth roots. Clin Oral Implants Res. 2017 Mar;28(3):334-340. doi: 10.1111/clr.12803. Epub 2016 Mar 29. PMID 27028526
- [Result] Schwarz F, Golubovic V, Becker K, Mihatovic I. Extracted tooth roots used for lateral alveolar ridge augmentation: a proof-of-concept study. J Clin Periodontol. 2016 Apr;43(4):345-53. doi: 10.1111/jcpe.12481. Epub 2016 Mar 17. PMID 26580310
- [Result] Schwarz F, Golubovic V, Mihatovic I, Becker J. Periodontally diseased tooth roots used for lateral alveolar ridge augmentation. A proof-of-concept study. J Clin Periodontol. 2016 Sep;43(9):797-803. doi: 10.1111/jcpe.12579. Epub 2016 Jun 25. PMID 27169909
- [Result] Becker K, Jandik K, Stauber M, Mihatovic I, Drescher D, Schwarz F. Microstructural volumetric analysis of lateral ridge augmentation using differently conditioned tooth roots. Clin Oral Investig. 2019 Jul;23(7):3063-3071. doi: 10.1007/s00784-018-2723-4. Epub 2018 Nov 9. PMID 30413950
- [Result] Schwarz F, Mihatovic I, Popal-Jensen I, Parvini P, Sader R. Influence of autoclavation on the efficacy of extracted tooth roots used for vertical alveolar ridge augmentation. J Clin Periodontol. 2019 Apr;46(4):502-509. doi: 10.1111/jcpe.13090. Epub 2019 Mar 28. PMID 30791121